CLINICAL TRIAL: NCT00192413
Title: A Prospective, Randomized, Open-Label, Controlled Trial to Compare the Safety, Tolerability, and Efficacy of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (CAIV-T) With Inactivated, Influenza Vaccine, Trivalent, Types A & B, in Adults Aged 60 Years and Older
Brief Title: Trial to Compare the Safety, Tolerability, and Efficacy of Influenza Virus Vaccine, (CAIV-T) With Inactivated, Influenza Vaccine, Trivalent, Types A & B, in Adults Aged 60 Years and Older Against Culture-confirmed Influenza
Acronym: FluMist
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Raburn Mallory, MD/ Sr Dir Clinical Development, MedImmune
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D153-P516
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold-adapted influenza vaccine trivalent (CAIV-T) (Experimental): A single 0.2 mL dose of 10^7 fluorescent focus units was administered intranasally.
  Interventions: Biological: Cold-adapted influenza vaccine trivalent (CAIV-T)
- Trivalent Inactivated Vaccine (TIV) (Active Comparator): A single dose was administered by intramuscular injection.
  Interventions: Biological: Trivalent Inactivated Vaccine (TIV)

INTERVENTIONS:
Biological: Cold-adapted influenza vaccine trivalent (CAIV-T) — Liquid CAIV-T vaccine for this study consisted of 3 cold-adapted, attenuated, reassortant strains, representing the HA and NA antigens of the A/New Caledonia/20/99 (H1N1), A/Panama/2007/99 (H3N2), and B/Victoria/504/2000 influenza strains. The vaccine contained no preservatives and had a pH of 7.2 ± 0.5.
  Other Names: FluMist
  Arms: Cold-adapted influenza vaccine trivalent (CAIV-T)
Biological: Trivalent Inactivated Vaccine (TIV) — Commercially available TIV, inactivated influenza vaccine (Split Virion) BP (Aventis Pasteur MSD, Lyon, France) was administered IM according to the manufacturer's dosing instructions (one 0.5-mL IM dose for adults).
  Arms: Trivalent Inactivated Vaccine (TIV)

SUMMARY:
To demonstrate that the efficacy over a defined surveillance period against culture-confirmed influenza-illness caused by community-acquired subtypes antigenically similar to those contained in the vaccine, in adults aged at least 60 years at enrollment, of a single intranasally (IN) -administered dose of a liquid formulation of influenza virus vaccine,(CAIV-T) is non inferior compared with that of a single dose of commercially available influenza vaccine inactivated (TIV) administered intramuscularly (IM) prior to the anticipated commencement of the influenza season.

ELIGIBILITY:
Inclusion Criteria:

* who are aged at least 60 years or older at the time of enrollment;
* who are determined by medical history, physical examination and clinical judgement to be eligible for this study;
* who have provided written informed consent after the nature of the study has been explained;
* who will be available for duration of the trial (from enrollment to November 30th, 2003);
* who can be reached by study staff for the post-vaccination and weekly surveillance contacts [telephone, clinic or home visit].

Exclusion Criteria:

* who are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* who are a resident of a nursing home or long-term care facility or other institution receiving skilled or semi-skilled nursing care (refer to Influenza study specific manual). An ambulatory subject who is a resident of a retirement home or village is eligible for the trial;
* with any signs of renal insufficiency requiring supportive therapy or progressive neurological disease. (Subjects with other stable pre-existing disease, defined as disease not requiring change in therapy or hospitalization within 12 weeks before receipt of study vaccination will be eligible).
* with evidence of dementia or other severe cognitive impairment based on Mini Mental State Examination (MMSE) scores (refer to Influenza study specific manual);
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids; or cytotoxic agents;
* who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* have an immunosuppressed or an immunocompromised individual living in the same household;
* with a documented history of hypersensitivity to egg or egg protein or any other component of the CAIV-T or TIV vaccine;
* who were administered any live virus vaccine within one month prior to vaccination or expected to receive another live virus vaccine within one month of vaccination in this study;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* who received a dose of influenza treatment (commercial or investigational) one month prior to enrollment. The prophylactic use of influenza antivirals is not permitted.
* who receive any influenza vaccine in the 6 months prior to enrollment, or intend to receive a non-study influenza vaccine after enrollment;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results; Note: A pregnant household member is not considered a contraindication to enrollment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3009 (Actual)
Dates: Start 2002-03; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
The first episode of a culture-confirmed influenza-illness, caused by community-acquired subtypes antigenically similar to those contained in the vaccine, which occurs at least 15 days following receipt of a dose of study vaccine. | Dosing through 30Nov2002
  The criteria for obtaining nasal and throat swabs for viral culture were any one of the following: A feeling of "feverishness", An oral temperature ≥37.2ºC, Sore throat, New or increased cough, Malaise, Myalgia. Swabs for viral cultures were also obtained, if, in the opinion of the investigator, the symptom complex so warranted.

SECONDARY OUTCOMES:
The first episode of a culture-confirmed influenza-illness, caused by any community-acquired subtype, which occurs at least 15 days following receipt of a dose of study vaccine. | 15 days after dosing through 30Nov2002
  The criteria for obtaining nasal and throat swabs for viral culture were any one of the following: A feeling of "feverishness", An oral temperature ≥37.2ºC, Sore throat, New or increased cough, Malaise, Myalgia. Swabs for viral cultures were also obtained, if, in the opinion of the investigator, the symptom complex so warranted.
The first episode in a study subject of a culture-confirmed influenza illness caused by community-acquired virus of each of the subtypes antigenically similar to those contained in the vaccine | 15 days after dosing through 30Nov2002
  The criteria for obtaining nasal and throat swabs for viral culture were any one of the following: A feeling of "feverishness", An oral temperature ≥37.2ºC, Sore throat, New or increased cough, Malaise, Myalgia. Swabs for viral cultures were also obtained, if, in the opinion of the investigator, the symptom complex so warranted.
The first episode in a study subject of a culture-confirmed influenza illness caused by any community-acquired virus of each of the subtypes. | 15 days after dosing through 30Nov2002
  The criteria for obtaining nasal and throat swabs for viral culture were any one of the following: A feeling of "feverishness", An oral temperature ≥37.2ºC, Sore throat, New or increased cough, Malaise, Myalgia. Swabs for viral cultures were also obtained, if, in the opinion of the investigator, the symptom complex so warranted.
The first episode of influenza-like illness | 15 days after dosing through 30Nov2002
Incidence of clinic visits | 15 days after dosing through 30Nov2002
  A possibility of multiple visits per subject; each visit will be counted once in the analysis.
Incidence of hospitalization | 15 days after dosing through 30Nov2002
Incidence of confirmed pneumonia | 15 days after dosing through 30Nov2002
  Pneumonia means one or more areas of acute interstitial or alveolar infiltrates documented radiographically
Incidence of death due to influenza-like illness | 15 days after dosing through 30Nov2002
  With or without confirmation by viral culture or PCR analysis
Incidence of seroconversion | Day 0-35
  Seroconversion is defined as at least a 4-fold increase in titer from baseline to the sample 35 plus or minus 7 days after vaccination. all subjects were to provide serum samples at 2 time points: at study visit 1 prior to vaccination with CAIV-T or TIV, and 35 days ± 7 days following vaccination (study visit 2).
Incidence of systemic reactogenicity events | Day 0-10
  The 12 systemic reactions were fever with 3 grades defined as ≥37.2°C, ≥38.6°C, and ≥40°C based on the temperature reported on the diary card in addition to the 9 events reported on the diary card.
Incidence of local reactions | Days 0-10
  The local reactions were pain, redness (2 grades: any and significant), and swelling (also 2 grades).
Incidence of adverse events | Days 0-10

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (4):
- South Africa (4):
  - Docnor House, Durban North, Dwazulu Natal
  - Hazelmed Family Practice, Hazelwood, Pretoria
  - Jansen van Rensburg, eManzimtoti
  - Christiaan Tertius de Villiers, Scottburgh South

REFERENCES:
- [Result] Forrest BD, Steele AD, Hiemstra L, Rappaport R, Ambrose CS, Gruber WC. A prospective, randomized, open-label trial comparing the safety and efficacy of trivalent live attenuated and inactivated influenza vaccines in adults 60 years of age and older. Vaccine. 2011 May 9;29(20):3633-9. doi: 10.1016/j.vaccine.2011.03.029. Epub 2011 Apr 5. PMID 21440036